CLINICAL TRIAL: NCT04202731
Title: Sleep, Insulin Sensitivity, and Weight in Adolescents Post-bariatric Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic impacted recruitment
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0926
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Extension (Experimental): Participants will be asked to extend their time in bed with the goal of improving the total time they sleep each night.
  Interventions: Behavioral: PBS Study

INTERVENTIONS:
Behavioral: PBS Study — Sleep extension intervention

SUMMARY:
Assessing sleep and circadian health in severely obese adolescents undergoing bariatric surgery and examine relation to health outcomes including insulin sensitivity and percent weight loss to date at 1-year and evaluate the impact of sleep extension on health outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

* ages 12-21 years
* attending high school or middle school (peak period for insufficient and delayed sleep)
* completion of bariatric surgery procedure (i.e., vertical sleeve gastrectomy) within the past 2 years but not less than 6 months prior to study participation
* All must also be Tanner Stage 5

Exclusion Criteria:

* regular use of medications affecting sleep (e.g., stimulants, atypical antipsychotics, melatonin or other sleep aids) or insulin resistance (systemic steroids, other oral diabetes medications)
* HbA1c ≥6.5%
* intelligence quotient (IQ) <70 or severe mental illness

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Sleep duration | 1 week
  Total sleep time at night in hours

CONTACTS AND LOCATIONS:
Overall Officials: Jill L Kaar, PhD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No